CLINICAL TRIAL: NCT03991897
Title: Nutritional Ketosis: a Novel Metabolic Strategy to Treat Lymphedema Patients?
Acronym: KETOLYMPH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S61767; 2018-002968-10 (EudraCT Number)
Record Dates: First submitted 2018-11-16; First posted 2019-06-19 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-08

CONDITIONS: Lymphedema; Ketogenic Dieting; Ketone Ester Supplement
Keywords: ketosis; lymphedema; dermal backflow
MeSH Terms: conditions — Lymphedema; Ketosis | interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: After baseline assessment, patients will be randomized in one of the treatment groups.
  Randomization is performed according to 'www.randomization.com'. This free generator randomizes each subject to a single treatment by using the method of randomly permuted blocks.
  Assessments are performed by a person blinded to the treatment allocation groups.
  Randomization will be stratified for baseline lymphedema volume (3-9.9%, 10.0-19.9% and ≥20%), and gender (females or males). The staff members who perform the measurements are blinded for the allocation.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ketogenic diet (Experimental): the intervention will consist of 3 phases: a two week run-in period, 12 weeks strict KD and 6 months Modified Atkins Diet.
  During the run-in period, patients will become familiar with their diet and, in particular, they will learn which foods are allowed and which are not. Ketogenic ratio wil build up to 3:1 - 4:1, ensuring protein needs.
  Interventions: Dietary Supplement: Ketogenic diet
- Isocaloric diet (Active Comparator): During the run-in period, the dietician will discuss the diet and maintenance of an isocaloric diet with the patients. As such, the diet of the control group will not change from their normal dietary pattern. In the latter case, the patient will be asked to change the diet to a normal Belgian diet, according to Flemisch dietary guidelines.
  Interventions: Dietary Supplement: Isocaloric diet
- Ketone ester supplementation (Experimental): Arm Description: the intervention will consist of 3 phases: a two week run-in period, 12 weeks strict of Ketone ester supplementation and 6 months of the follow-up with a healthy diet. Ke supplements will be ingested 3 times a day separately from a meal in fixed doses of 25g. If blood β-OHB levels are substantially below 3mmol/L, a weight-based dosing of the KEs (up to 0.5g/kg bodyweight), rather than a fixed dosing strategy, will be utilized.
  Interventions: Dietary Supplement: Ketone ester supplementation

INTERVENTIONS:
Dietary Supplement: Ketogenic diet — Multivit and Metarelax. This multivitamin and Magnesium supplement will provide necessary vitamins and decrease ketone-flu sympotms, repsectively.
  Arms: Ketogenic diet
Dietary Supplement: Isocaloric diet — Patients will follow an isocaloric diet
  Arms: Isocaloric diet
Dietary Supplement: Ketone ester supplementation — 25g of a ketone monoester, ingested 3 times a day for a period of 12 weeks. Ingestion is separated from a meal and interspersed by at least 4 hours to ensure maximal available ketone bodies circulating in the blood.
  Arms: Ketone ester supplementation

SUMMARY:
Lymphedema is a debilitating disorder that severely impairs the quality of life of the patients and requires life-long attention. Treatment for lymphatic dysfunction remains largely symptomatic, without real cure. According to the International Society of Lymphology, lymphedema has to be treated with Decongestive Lymphatic Therapy.

Research in the lab of Angiogenesis and Vascular Metabolism (PCA lab) reported in mice that metabolism of endothelial cells controls vessel sprouting. Experiments showed that a ketogenic diet (KD) reduced the edema of the mice tail and enhanced the lymphatic transport. Based on these proof-of-concept data, the investigators plan to test this innovative concept to ameliorate lymph vessel dysfunction in lymphedema patients. Randomisation will be performed between a ketogenic diet and an isocaloric diet with and without ketone ester supplementation.

DETAILED DESCRIPTION:
Lymphedema is a debilitating disorder that severely impairs the quality of life of the patients and requires life-long attention. It can be classified as primary or secondary, based on the etiology. Primary lymphedema is a rare, congenital disorder caused by inherited genetic mutation on a number of genes that are essential for lymphatic vessel development and function. Acquired (or secondary) lymphedema is a consequence of lymphatic trauma, predominantly due to surgery or radiotherapy for various types of cancers, with axillary and/or inguinal lymph node dissection being the most common cause. At the cellular level, perturbed or dysfunctional lymphatic drainage triggers accumulation of interstitial fluid, negatively affects cellular behavior, and induces infiltration of fibroblasts, adipocytes and keratinocytes, eventually leading to possible fibrosis and ulceration.

Upper extremity lymphedema most commonly affects breast cancer patients, while lower extremity lymphedema is typically associated with gynecological cancers, prostate cancer, lymphoma and melanoma. Besides the functional impairments, lymphedema severely reduces the quality of life, causing psychosocial problems such as depression, sexual dysfunctions, social avoidance and a decrease in self-confidence. While the prevalence of lymphedema is relatively high (1.33-1.44 pro mille), its true prevalence is likely underestimated and 1 in 6 patients undergoing treatment for a solid tumor ultimately develops lymphedema.

Nevertheless, treatment for lymphatic dysfunction remains largely symptomatic, without real cure. According to the International Society of Lymphology, lymphedema has to be treated with Decongestive Lymphatic Therapy, a two-stage treatment program. During the first or intensive phase, lymphedema has to be maximally reduced: this phase consists of skin care, manual lymph drainage (MLD), multi-layer bandaging and exercise therapy. The second or maintenance phase aims to conserve and optimize the result obtained in the first phase, and consists of skin care, compression by a low-stretch elastic sleeve, exercises and MLD. Skin care, multi-layer bandaging, elastic sleeve and exercises are treatment modalities that can be performed by the patients themselves, after careful instruction from the physician. On the contrary, MLD has to be applied by a physical therapist and hence entails a big financial cost for the patient and the Health Care. In addition, reductive techniques, such as direct excision and liposuction, can be applied to patients with more advanced stages of lymphedema with a predominant fibrofatty component. Encouraging initial results, i.e. symptomatic improvement and reduction in excess volume, have been obtained with lymphovenous bypass, the microsurgical anastomosis of collecting lymphatic vessels to adjacent venules, and vascularized lymph node transplantation, where lymph nodes are harvested from an unaffected region and transferred to the lymphedematous area. However, all the treatments available so far can offer only stabilisation of lymphedema and prevent further evolution, but they do not offer a definitive cure. There is thus a large unmet need to develop new effective therapies for lymphedema and, more general, lymph vessel dysfunction. In contrast to various strategies inhibiting lymphatic vessel growth, stimulating lymphatic vessel growth has been more challenging; there is currently no approved clinical strategy for ameliorating lymphatic dysfunctions. In this trial we will evaluate an entirely novel pro-lymphangiogenic strategy, not based on the delivery of lymphangiogenic growth factors, but rather based on modulating lymphatic endothelial cell metabolism. The lab of Angiogenesis and Vascular Metabolism (PCA lab), Catholic University Leuven, led by Prof. Peter Carmeliet recently reported that metabolism (glycolysis, fatty acid β-oxidation, glutamine metabolism) of endothelial cells, the cells lining blood vessels, controls vessel sprouting. Initial experiments from this PCA lab indicate that the Ketogenic Diet (KD) , which is effective in increasing the levels of ßOHB both in the plasma and lymph, ameliorates the disease outcome in the mouse (tail) model of lymphedema, by reducing edema formation over time. Strikingly, lymphangiography with Evans blue dye revealed that KD improves lymph vessel function, increasing dye uptake after subcutaneous injection in the lymphedematous tissue and its drainage into lymph, plasma and lymph nodes.

Based on these proof-of-concept data, the investigators plan to test this innovative concept to ameliorate lymph vessel dysfunction in lymphedema patients.

Randomisation will be performed between 3 arms: a ketogenic diet and a isocaloric diet without or including ketone monoester supplementation (KE).

After randomization and baseline measurements (determination of energy requirements and intake), the intervention will consist of 3 phases: a two week run-in period, 12 weeks of strict KD or KE and a 6 months Modified Atkins Diet or an isocaloric diet. The first phase, the two week run-in period, is the establishment of the individual ketosis level (on average after five days ketosis is introduced). During this run-in period, the exact ratio of lipids over proteins and carbohydrates will be determined per patient based on an isocaloric diet; this ratio will vary per patient and over time. During this run-in period, patients will become familiar with their diet, and in particular, they will learn which foods are allowed and which are not. To assist the patients, the ketobel program (a computer program developed by the metabolic dieticians of the Clinical Nutrition Unit, University Hospital Leuven) will allow the calculation of the exact amount of foods/lipids each patient can/needs to consume. The instructions given by the program will allow patients to create a menu according to their personal preferences, with the final aim of increasing the adherence to the KD. A dietician will assist every participant intensively in this run-in period (10 h/week). To ensure ketotic state, ketosis will be measured twice a day (morning and evening) using urinary sticks. If there is a change in the ketotic state for the KD, the lipid/non-lipid fraction ratio will be adjusted in collaboration with the dietician.

The KE group will include ketone esters within their dietary intake. Fixed doses of 25g will be consumed 3 times a day. Ingestion will be detached from a meal, with at least 4-hour intervals in between doses to induce 12 hours of ketosis. If blood β-OHB levels are substantially below 3mmol/L, a weight-based dosing of the KEs (up to 0.5g/kg bodyweight), rather than a fixed dosing strategy, will be utilized.

In the second phase, the patients following the KD for 12 weeks the dietician will assist the patient during this phase 2 hours/week. This support is necessary as the lipid/non-lipid ratio to obtain ketosis varies over time as well. The KE group will adhere to an isocaloric healthy diet including 3 doses of 25g of ketone esters daily. A researcher will assess on a weekly basis general health status, body parameters (weight, waist circumference), physical activity, weight loss and compliance to diet. The plasma metabolite profile (different types of cholesterol, triglycerides, fasting glucose, hsCRP, ketone bodies) will be performed every 3 weeks. To stimulate adherence to the diet, chat sessions will be organized between patients and a dietician, as moderator; these sessions will take place once a week and allow patients to exchange ideas/recipes about the diet and to motivate each other. These chat sessions have been organized previously by the members of the Clinical and Experimental Endocrinology group in other projects and were considered by the patients as an added value and a stimulation to continue with the intervention.

In the third phase, the patients' diet will be less strict and adapted to a Modified Atkins Diet. This shift is necessary to enhance adherence on the one hand and to allow follow-up for a longer period.

ELIGIBILITY:
Inclusion Criteria:

* >18 years;
* unilateral lymphedema of the arm lymph node dissection
* lymphedema onset less than a year before the therapy starts
* lymphedema defined as >3% volume difference between both arms
* lymphedema stage 1, stage 2a or stage 2b
* absence of pregnancy at the time of enrollment and willingness to use adequate contraceptive measures until the end of the study;
* oral and written approval of the informed consent presented at the time of the consultation by the physicians;
* understanding Dutch

Exclusion Criteria:

* <18 years;
* edema of the limb with different etiology or later stage/onset as specified in the inclusion criteria;
* presence of active cancer
* pregnancy or active breastfeeding;
* impossibility to participate for the entire study period;
* mentally or physically unable to participate to the study;
* presence of gastrointestinal intolerance or other serious illness (e.g. renal failure, hepatic dysfunction, heart failure, neurological impairment);
* presence of diabetes or other metabolic disease;
* contra-indication for the use of indocyanine green (ICG): allergy to ICG or iodine, hyperthyroidism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in lymphatic transport | Up to 12 weeks
  Measured with lymphoscintigraphy
Change in lymphatic transport | up to 12 weeks
  Measured by lymphofluoroscopy

SECONDARY OUTCOMES:
Change in edema volume | 12 weeks
  Measured with tape circumference
Change in edema volume | 12 weeks
  measured with volumeter
Changed quality of life | 12 weeks
  measured with Lymph ICF (international classification of functioning, disability and Health), a scale from 0-10 on 29 items, total score ranged from 0-100, 0-4: indicate no problem; 5-24 a small problem; 26-49: moderate problem; 50-95: severe problem; 96-100: very severe problem
Lymphatic function at 6 months | 6 months
  Change in dermal backflow score at 6-month follow-up
Change in edema volume at 6 months | up to 6 months
  measured with volumeter
Change in edema volume at 6 months | up to 6 months
  measured with tape circumference
Changed quality of life after 6 months | 6 months
  measured with Lymph ICF (international classification of functioning, disability and Health), a scale from 0-10 on 29 items, total score ranged from 0-100, 0-4: indicate no problem; 5-24 a small problem; 26-49: moderate problem; 50-95: severe problem; 96-100: very severe problem

OTHER OUTCOMES:
Cost-effectiveness | up to 6 months
  Difference in cost-effectiveness between nutritional ketosis, induced by either consumption of a CKD or ingestion of KE supplements, and a healthy diet at 6-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Timmermans, Msc, Principal Investigator — KU Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lodewijckx I, Matthys C, Verheijen J, Verscuren R, Devoogdt N, Van der Schueren B, Goffin K, Fourneau I, Thomis S. Potential therapeutic effect of a ketogenic diet for the treatment of lymphoedema: Results of an exploratory study. J Hum Nutr Diet. 2024 Aug;37(4):885-891. doi: 10.1111/jhn.13330. Epub 2024 Jun 4. PMID 38837503
- [Result] Garcia-Caballero M, Zecchin A, Souffreau J, Truong AK, Teuwen LA, Vermaelen W, Martin-Perez R, de Zeeuw P, Bouche A, Vinckier S, Cornelissen I, Eelen G, Ghesquiere B, Mazzone M, Dewerchin M, Carmeliet P. Role and therapeutic potential of dietary ketone bodies in lymph vessel growth. Nat Metab. 2019 Jul;1(7):666-675. doi: 10.1038/s42255-019-0087-y. Epub 2019 Jul 12. PMID 32694649